CLINICAL TRIAL: NCT04314024
Title: Phase I, Randomized, Open-Label, Single-Dose, Three Period, Six-Sequence Crossover Study to Determine the Relative Bioavailability of the Evobrutinib Intended Commercial Tablet Formulation (TF2) Compared to the Clinical Tablet Formulation (TF1) and Evaluate the Effect of Food on TF2 Bioavailability in Healthy Participants
Brief Title: Relative Bioavailability (rBA) of Evobrutinib Intended Commercial and Clinical Tablets, and Effect of Food on Intended Commercial Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200527_0077; 2019-004738-40 (EudraCT Number)
Record Dates: First submitted 2020-03-17; First posted 2020-03-18 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: Evobrutinib; Pharmacokinetics; Relative Bioavailability; Crossover
MeSH Terms: interventions — evobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Evobrutinib: Treatment Sequence 1: A-B-C (Experimental): Participants will receive single oral dose of TF1 (Treatment A) evobrutinib on Day 1 under fasted condition in period 1, followed by single oral dose of TF2 (Treatment B) on Day 3 under fasted condition in period 2, followed by TF2 (Treatment C) on Day 5 under fed condition in period 3. There will be 48 hours washout period between each treatment period.
  Interventions: Drug: Evobrutinib
- Evobrutinib: Treatment Sequence 2: A-C-B (Experimental): Participants will receive single oral dose of TF1 (Treatment A) evobrutinib on Day 1 under fasted condition in period 1, followed by TF2 (Treatment C) on Day 3 under fed condition in period 2, followed by single oral dose of TF2 (Treatment B) on Day 5 under fasted condition in period 3. There will be 48 hours washout period between each treatment period.
  Interventions: Drug: Evobrutinib
- Evobrutinib: Treatment Sequence 3: B-A-C (Experimental): Participants will receive single oral dose of TF2 (Treatment B) on Day 1 under fasted condition in period 1, followed by single oral dose of TF1 (Treatment A) evobrutinib on Day 3 under fasted condition in period 2, followed by TF2 (Treatment C) on Day 5 under fed condition in period 3. There will be 48 hours washout period between each treatment period.
  Interventions: Drug: Evobrutinib
- Evobrutinib: Treatment Sequence 4: B-C-A (Experimental): Participants will receive single oral dose of TF2 (Treatment B) on Day 1 under fasted condition in period 1, followed by TF2 (Treatment C) on Day 3 under fed condition in period 2, followed by single oral dose of TF1 (Treatment A) evobrutinib on Day 5 under fasted condition in period 3. There will be 48 hours washout period between each treatment period.
  Interventions: Drug: Evobrutinib
- Evobrutinib: Treatment Sequence 5: C-A-B (Experimental): Participants will receive single oral dose of TF2 (Treatment C) on Day 1 under fed condition in period 1, followed by single oral dose of TF1 (Treatment A) evobrutinib on Day 3 under fasted condition in period 2, followed by single oral dose of TF2 (Treatment B) on Day 5 under fasted condition in period 3. There will be 48 hours washout period between each treatment period.
  Interventions: Drug: Evobrutinib
- Evobrutinib: Treatment Sequence 6: C-B-A (Experimental): Participants will receive single oral dose of TF2 (Treatment C) on Day 1 under fed condition in period 1, followed by single oral dose of TF2 (Treatment B) on Day 3 under fasted condition in period 2, followed by single oral dose of TF1 (Treatment A) evobrutinib on Day 5 under fasted condition in period 3. There will be 48 hours washout period between each treatment period.
  Interventions: Drug: Evobrutinib

INTERVENTIONS:
Drug: Evobrutinib — Participants will receive single oral dose of evobrutinib either after an overnight fast of at least 10 hours (Treatment A and Treatment B), or under fed conditions that is within 30 minutes after start of high-fat meal (Treatment C) in period 1, 2 and 3.
  Other Names: M2951

SUMMARY:
The study will evaluate the relative bioavailability (rBA) of the intended commercial tablet formulation (Test Treatment, TF2) of Evobrutinib compared to the clinical tablet formulation (Reference Treatment, TF1) of Evobrutinib and to assess the effect of food on the bioavailability of the intended commercial tablet formulation of Evobrutinib.

ELIGIBILITY:
Inclusion Criteria:

* Participants are overtly healthy as medical evaluation, including no clinically significant abnormality identified on physical examination or laboratory evaluation and no active clinically significant disorder, condition, infection or disease that would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion
* Male or female participants agree to be consistent with local regulations on contraception methods
* Female participants are not pregnant or breastfeeding, and at least one of the following condition applies:
* Not a WOCBP or
* If a WOCBP, use a highly effective contraceptive method (that is, with a failure rate of <1 percent per year, preferably with low user dependency for the following time period:
* Before the first dose of the study intervention, if using hormonal contraception:
* Has completed at least one 4-week cycle of an oral contraception pill and either had or has begun her menses or
* Has used a depot contraceptive or extended-cycle oral contraceptive for least 28 days and has a documented negative pregnancy test using a highly sensitive assay and
* A barrier method
* During the intervention period
* After the study intervention period (that is after the last dose of study intervention is administered) for at least 90 days, plus 30 days (a menstrual cycle) after the last dose of study intervention and agree not to donate eggs (ova, oocytes) for reproduction during this period. The Investigator evaluates the effectiveness of the contraceptive method in relationship to the first dose of study intervention
* Females have a negative serum pregnancy test at the Screening Visit and within 24 hours before the first dose of study intervention
* The Investigator reviews the medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a female with an early undetected pregnancy
* Participants are stable non-smokers for at least 3 months preceding screening
* Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* History or presence of clinically relevant respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders.
* Prior history of cholecystectomy or splenectomy, and any clinically relevant surgery within 6 months prior to screening
* History of any malignancy
* History of chronic or recurrent acute infection or any bacterial, viral, parasitic or fungal infections within 30 days prior to screening and at any time between screening and admission, or hospitalization due to infection within 6 months prior to screening
* History of shingles within 12 months prior to screening
* History of drug hypersensitivity, ascertained or presumptive allergy/hypersensitivity to the active drug substance and/or formulation ingredients
* History of alcoholism or drug abuse within 2 years prior to screening, or evidence of such abuse as indicated by the laboratory assays conducted during screening
* History of residential exposure to tuberculosis, or a positive QuantiFERON® test within 4 weeks prior to screening
* Administration of live vaccines or live-attenuated virus vaccines within 3 months prior to screening
* Any condition, including findings in the laboratory tests, medical history, or other screening assessments, that in the opinion of the Investigator constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study's objectives, conduct, or evaluation
* Other protocol defined exclusion criteria could apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of Evobrutinib Under Fasted Conditions | Pre-dose up to 24 hours post-dose on Day 6
Area Under the Plasma Concentration-Time Curve from Time Zero to Infinity (AUC0-inf) of Evobrutinib Under Fasted Conditions | Pre-dose up to 24 hours post-dose on Day 6
Maximum Observed Plasma Concentration (Cmax) of Evobrutinib Under Fasted Conditions | Pre-dose up to 24 hours post-dose on Day 6
Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of Evobrutinib Under Fed Conditions | Pre-dose up to 24 hours post-dose on Day 6
Area Under the Plasma Concentration-Time Curve from Time Zero to Infinity (AUC0-inf) of Evobrutinib Under Fed Conditions | Pre-dose up to 24 hours post-dose on Day 6
Maximum Observed Plasma Concentration (Cmax) of Evobrutinib Under Fed Conditions | Pre-dose up to 24 hours post-dose on Day 6

SECONDARY OUTCOMES:
Number of Participants With Treatment -Emergent Adverse Events (TEAEs) Based on Severity Under Fasted Conditions | Day 1 up to Day 6
Number of Participants With Clinically Significant Change From Baseline in Vital Signs, Laboratory Parameters and Electrocardiogram Findings Under Fasted Conditions | Day 1 up to Day 6
  Number of participants with clinically significant change from baseline in vital signs, laboratory parameters and electrocardiogram findings will be reported
Area Under the Plasma Concentration-Time Curve From Time Zero to Time 24 Hours After Evobrutinib Administration (AUC0-24) | Pre-dose up to 24 hours post-dose on Day 6
Area Under The Plasma Concentration-Time Curve From Time Zero to Time 12 Hours After Evobrutinib Administration (AUC0-12) | Pre-dose up to 12 hours post-dose on Day 6
Time to Reach Maximum Plasma Concentration (Tmax) of Evobrutinib | Pre-dose up to 24 hours post-dose on Day 6
Time Prior to the First Measurable (non-zero) Concentration (t lag) of Evobrutinib | Pre-dose up to 24 hours post-dose on Day 6
Terminal First Order (elimination) Rate Constant (λz) of Evobrutinib | Pre-dose up to 24 hours post-dose on Day 6
Apparent Elimination Half Life (t1/2) of Evobrutinib | Pre-dose up to 24 hours post-dose on Day 6
Apparent Total Body Clearance (CL/f) of Evobrutinib | Pre-dose up to 24 hours post-dose on Day 6
Apparent Volume of Distribution During Terminal Phase (VZ/f) of Evobrutinib | Pre-dose up to 24 hours post-dose on Day 6
Relative Bioavailability of Test Treatment in Relation to Reference Treatment (Frel) | Pre-dose up to 24 hours post-dose on Day 6

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany, will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.merckgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200527_0077
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html